CLINICAL TRIAL: NCT03697746
Title: Comparison of Dexketoprofen, Paracetamol and Ibuprofen in the Treatment of Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, seçkin çiftçioğlu, Emergency Medicine, Pamukkale University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Pamukkkale University
Record Dates: First submitted 2018-09-30; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Acetaminophen; dexketoprofen trometamol; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paracetamol (Active Comparator): 1000 mg Paracetamol vial intravenously
  Interventions: Drug: paracetamol
- Dexketoprofen Trometamol (Active Comparator): 50 mg Dexketoprofen Trometamol vial intravenously
  Interventions: Drug: Dexketoprofen Trometamol
- Ibuprofen (Active Comparator): 400 mg Ibuprofen vial intravenously
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: paracetamol — paracetamol 1000 mg vial
  Other Names: Parol 1000 mg vial--Mefar medicine-İstanbul
  Arms: Paracetamol
Drug: Dexketoprofen Trometamol — dexketoprofen trometamol 50 mg bulb
  Other Names: Dexiren 50 mg bulb-İlko medicine-İdol
  Arms: Dexketoprofen Trometamol
Drug: Ibuprofen — ıbuprofen 400 mg vial
  Other Names: İntrafen 400mg/4ml flakon-Gen medicine- Ankara
  Arms: Ibuprofen

SUMMARY:
Our study will be performed on 300 patients who meet the criteria for joining the emergency service with primary dysmenorrhea.

3 drugs we will use: 1000 mg vial of paracetamol, dexketoprofen trometamol will be 50 mg ampoule and ibuprofen 400 mg vial

According to the visual analog scale and visual visual scale, we will ask the patient to rate her pain between 0 (no pain) and 10 (the most severe pain of her life).

We aim to determine the superiority of the drugs in passing the pain randomly by giving the 3 drugs that we mentioned to patients with pain above 5.

DETAILED DESCRIPTION:
Our research will be carried out in Pamukkale University Faculty of Medicine Department of Emergency Medicine in 12 months period. There will be a research assistant and / or a faculty member who will control the research for 24 hours in our emergency department with approximately 110000 adult patients / year.

Study criteria: Female patients with primary dysmenorrhea (abdomino-pelvic pain) in the 18-45 age range. The onset of symptoms should usually be a few hours - 1 day before the onset of visible vaginal bleeding. Possible systemic symptoms such as nausea, vomiting, diarrhea, headache, fatigue, irritability, and dizziness are also questioned and recorded in the data form. Patients with a Visual Analog Scale > 5 and those who require or are recommended nonsteroid antiinflammatory treatment.Patients who come with dysmenorrhea will be randomly selected and will be divided into three groups according to the pre-planned drug administration.

Group 1; Paracetamol 1000 mg Group 2; Dexketoprofen Trometamol 50mg Group 3; Ibuprofen 400 mg In the form of group to be administered intravenously. In case of unresponsiveness to treatment, intravenous Tramadol hcl 100mg will be administered after 45 minutes.

Pain scores of patients will be recorded using the Visual Analog Scale, 0-10 cm Visual Analog Scale, to score the degree of pain.During the process, O2 saturation monitorization, automatic manometer (blood pressure), rhythm monitorization (speed and rhythm) will be provided and all other medications during the operation will be recorded.

Pain scores will be recorded at 0, 15, 30, 45 and 60 minutes. In addition, heart rate, systolic blood pressure, diastolic blood pressure, respiration rate and O2 saturation (SPO2) will be recorded at 0, 15, 30, 60 minutes.

In addition, any side effects that may occur are recorded in the data sheet. If side effects are necessary, treatment will be applied. All information will be saved to the created work form

ELIGIBILITY:
Inclusion Criteria:

* Female patients with primary dysmenorrhea (abdomino-pelvic pain) between the ages of 18-45.
* The onset of symptoms should usually be a few hours - 1 day before the onset of visible vaginal bleeding.
* Possible systemic symptoms such as nausea, vomiting, diarrhea, headache, fatigue, irritability, and dizziness are also questioned and recorded in the data form.
* Patients with visual analogue scale score> 5 and those who need or need nonsteroidal anti-inflammatory treatment.

Exclusion Criteria:

* Severe liver, kidney and heart failure; asthma, nasal polyp, angioedema and urticaria against aspirin or other nonsteroidal antiinflammatory drugs;
* Active peptic ulcer, bleeding or perforation; to have a history of upper gastrointestinal disease;
* Patients with phenylketonuria;
* During pregnancy and lactation;
* Have asthma;
* Have taken analgesics in the last 4 hours;
* The age of pregnancy and not using birth control method; digoxin, lithium, furosemide and other diuretics, acetylsalicylic acid and coumarin group using anticoagulants and physical examination of the suspicion of acute abdomen and signs of peritoneal irritation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
ıtem pain intensity measure | 1 hour
  the patient will be given medication and will be asked to score between 0 and 10 on a visual analog scale.(0=no pain, 10= pain as bad as can be) every 15 minutes within 1 hour
ıtem pain intensity measure | 15 minute
  100 mg of tramadol hcl will be given when the patient's pain does not fall below 5 points on a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: SEÇKİN ÇİFTÇİOĞLU, Principal Investigator — PAMUKKALE UNİVERSİTY HOSPİTAL EMERGENCY MEDİCİNE
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data will be available within 1 year of study completion
Access Criteria: data access requests will be reviewed by on external independent review panel requestors will be required to sign a data access agreement

REFERENCES:
- [Background] Letzel H, Megard Y, Lamarca R, Raber A, Fortea J. The efficacy and safety of aceclofenac versus placebo and naproxen in women with primary dysmenorrhoea. Eur J Obstet Gynecol Reprod Biol. 2006 Dec;129(2):162-8. doi: 10.1016/j.ejogrb.2006.01.004. Epub 2006 May 3. PMID 16675091
- [Background] Ayan M, Tas U, Sogut E, Arici S, Karaman S, Esen M, Demirturk F. [Comparing efficiencies of diclofenac sodium and paracetamol in patients with primary dysmenorrhea pain by using Visual Analog Scale]. Agri. 2013;25(2):78-82. doi: 10.5505/agri.2013.42103. Turkish. PMID 23720082
- [Background] Iacovides S, Baker FC, Avidon I. The 24-h progression of menstrual pain in women with primary dysmenorrhea when given diclofenac potassium: a randomized, double-blinded, placebo-controlled crossover study. Arch Gynecol Obstet. 2014 May;289(5):993-1002. doi: 10.1007/s00404-013-3073-8. Epub 2013 Nov 5. PMID 24190696